CLINICAL TRIAL: NCT06301958
Title: The Effects and Molecular Mechanisms of Dextrose Prolotherapy on Articular Cartilage
Brief Title: Dextrose Prolotherapy on Articular Cartilage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, HSU, HUNG-CHIH, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202102567A3
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Arthritis Knee
Keywords: Dextrose; Prolotherapy; Joint Pain; Synovial Fluid
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dextrose prolotherapy (Experimental): A subject received a single intra-articular injection of 25% hypertonic glucose solution 10 mL (1:1 of 50% dextrose and normal saline) into one knee with arthritis after aspiration of all synovial fluid.
  Interventions: Drug: Dextrose prolotherapy

INTERVENTIONS:
Drug: Dextrose prolotherapy — A 25% dextrose solution is used to relieve arthritis of the knee joint like osteoarthritis and rheumatoid arthritis.
  Other Names: Regenerative injection therapy

SUMMARY:
Dextrose prolotherapy is a controversial injection therapy in sports medicine. Currently, 25% hypertonic glucose solution is commonly used in clinical practice. Although this method has a certain therapeutic effect, there is still some controversy about the molecular mechanism of dextrose prolotherapy. In the past, it was thought that local stimulation would increase inflammatory reactions such as local leukocyte and macrophage infiltration and restart the "self-healing mechanism." However, some studies have pointed out that this treatment can cause cell apoptosis. In my clinical work, I often perform dextrose prolotherapy. I deeply feel the importance of exploring the detailed mechanism of action of this therapy in order to apply this therapy more appropriately to patients. We believe that the concentration of 25% hypertonic glucose solution should show a stepwise decrease in the joint cavity. Our preliminary cell experiment results using 2-fold serial dilutions of 25% glucose solution showed that 25%, 12% and 6% glucose solution will trigger the apoptosis of chondrocytes, vascular endothelial cells and immune cells, and will also inhibit the expression of the pro-inflammatory factor IL-6. Glucose solution below 3% will not have the effect of inducing apoptosis on cells. We believe that the therapeutic effect of 25% hypertonic glucose solution in the joint cavity may have cell-specific effects as the concentration changes dynamically. Therefore, in this study, we will clarify the therapeutic mechanism of dextrose prolotherapy for arthritis through basic research and clinical specimen analysis. The clinical research part will use clinical synovial fluid specimens to verify the therapeutic mechanism of hypertonic glucose dissolution. The joint pain level assessment of different types of patients (OA and RA) before dextrose prolotherapy (preliminary period), 1 month after treatment (midterm period) and 3 months after treatment (late period) will be collected, and joint effusion will be measured. Further analyze the cell apoptosis and concentration changes of inflammatory response factors in the liquid.

We hope that through this study, we will have a clear understanding of the molecular mechanism of dextrose prolotherapy on joint component cells. This result will have reference value for the more appropriate application of dextrose prolotherapy in the treatment of human cartilage-related lesions.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a written consent form
* Adult men and women with arthritis

Exclusion Criteria:

* Pregnant or lactating women
* Septic arthritis
* Those who have undergone joint surgery within 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline, 1 month after treatment, and 3 months after treatment
  Measurement of knee pain

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | baseline, 1 month after treatment, and 3 months after treatment
  Osteoarthritis Index
Interleukin 6 (IL-6) | baseline, 1 month after treatment, and 3 months after treatment
  An inflammation-related biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chih Hsu, PhD, Principal Investigator — Chang Gung Memorial Hospital, Chiayi
Locations (1):
- Chang Gung Memorial Hospital, Chiayi, Chiayi City, 嘉義市, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing upon request